CLINICAL TRIAL: NCT00912028
Title: Multicenter, Single-masked, Randomized, Parallel, Controlled Study to Compare Senofilcon A Contact Lenses to Currently Used Contact Lenses
Brief Title: Clinical Performance Comparison of Several Different Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOH--BRA-001
Record Dates: First submitted 2009-05-29; First posted 2009-06-03 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- senofilcon A (Active Comparator): contact lens
  Interventions: Device: senofilcon A
- lotrafilcon B (Active Comparator): contact lens
  Interventions: Device: lotrafilcon B
- balafilcon A (Active Comparator): contact lens
  Interventions: Device: balafilcon A
- methafilcon A (Active Comparator): contact lens
  Interventions: Device: methafilcon A
- vifilcon A (Active Comparator): contact lens
  Interventions: Device: vifilcon A

INTERVENTIONS:
Device: senofilcon A — contact lens
  Arms: senofilcon A
Device: lotrafilcon B — contact lens
  Arms: lotrafilcon B
Device: balafilcon A — contact lens
  Arms: balafilcon A
Device: methafilcon A — contact lens
  Arms: methafilcon A
Device: vifilcon A — contact lens
  Arms: vifilcon A

SUMMARY:
The purpose of the study is to evaluate the possible benefits of second generation silicone hydrogel contact lenses.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* be existing soft contact lens wearers of the study control lenses
* require a distance visual correction in both eyes
* have a contact lens spherical distance requirement between -1.00 diopters (D) and -8.00D in both eyes
* have astigmatism less than or equal to 1.00D in both eyes
* be able to wear lenses available for this study
* be corrected to a visual acuity of 6/9 (20/30) or better in each eye
* have normal eyes with no evidence of abnormality or disease

Exclusion Criteria:

Subject are excluded for the following reasons:

* monovision corrected
* worn lenses extended wear in the last 3 months.
* require concurrent ocular medication
* grade 3 or 4 abnormalities
* grade 3 corneal staining in more than two regions
* anterior ocular surgery
* any other ocular surgery or injury within 8 weeks prior to study enrollment
* abnormal lachrymal secretions
* pre-existing ocular irritation that would preclude contact lens fitting
* corneal irregularities
* Polymethyl methacrylate (PMMA) or Rigid Gas Permeable (RGP) lens wear in past 12 weeks
* any systemic illness which would preclude contact lens wear
* diabetes
* infectious or immunosuppressive disease
* pregnancy or lactating, or planning pregnancy at time or enrollment
* participating in a concurrent clinical study or within last 60 days
* allergy to the standardized study care solution

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2010-02-01 (Actual); Study Completion 2010-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Leite Arieta, MD, PhD, Principal Investigator — Associate Professor - Ophthalmolgy, University of Campinas, Brazil
Locations (9):
- Brazil (9):
  - Salvador, Estado de Bahia
  - Maringá, Paraná
  - Recife, Pernambuco
  - Rio de Janeiro, Rio de Janeiro
  - Campinas, São Paulo
  - Marília, São Paulo
  - Ribeirão Preto, São Paulo
  - Santo André, São Paulo
  - São Paulo, São Paulo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Senofilcon A | Lotrafilcon B | Balafilcon A | Methafilcon A | Vifilcon A
Started | 35 | 3 | 13 | 17 | 3
Completed | 30 | 0 | 13 | 16 | 0
Not Completed | 5 | 3 | 0 | 1 | 3
Not completed — Lost to Follow-up | 2 | 3 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This population includes those who were qualified to be in the analysis population. Demographics are not available for those who were excluded or discontinued.
Groups:
- Total: Total of all reporting groups
Arm/Group | Senofilcon A | Balafilcon A | Methafilcon A | Total
Number analyzed (Participants) | 30 | 13 | 16 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (3.9) | 22.7 (3.5) | 27.0 (4.2) | 24.5 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 7 | 13 | 46
  Male | 4 | 6 | 3 | 13
Region of Enrollment [Number; unit: participants]
  Brazil | 30 | 13 | 16 | 59

OUTCOME MEASURES:

1. Primary Outcome: Limbal Hyperemia (Redness)
Description: Subject distribution according to limbal hyperemia scale in each eye during the 2-week Follow-up Visit. For this scale, 0 is lowest and 4 is greatest. If present in at least one eye, then it is counted.
Time Frame: 2 weeks
Population: Analysis is on those subjects who were enrolled, randomized, and completed the study.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Senofilcon A | Balafilcon A | Methafilcon A
Number analyzed (Participants) | 30 | 13 | 16
Number analyzed (eyes) | 60 | 26 | 32
eyes
  Grade 0 | 40 | 14 | 24
  Grade 1 | 12 | 4 | 4
  Grade 2 | 8 | 8 | 4
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

2. Primary Outcome: Limbal Hyperemia (Redness)
Description: Subject distribution according to limbal hyperemia scale in each eye during the 4-week Follow-up Visit. For this scale, 0 is lowest and 4 is greatest. If present in at least one eye, then it is counted.
Time Frame: 4 weeks
Population: Analysis is on those subjects who are enrolled, randomized to a study arm, and who completed the study.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Senofilcon A | Balafilcon A | Methafilcon A
Number analyzed (Participants) | 30 | 13 | 16
Number analyzed (eyes) | 60 | 26 | 32
eyes
  Grade 0 | 46 | 16 | 18
  Grade 1 | 10 | 4 | 12
  Grade 2 | 6 | 4 | 2
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

3. Primary Outcome: Bulbar Hyperemia (Redness)
Description: Subject distribution according to bulbar hyperemia scale in each eye during the 2-week Follow-up Visit. For this scale, 0 is lowest and 4 is greatest. If present in at least one eye, then it is counted.
Time Frame: 2 weeks
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Senofilcon A | Balafilcon A | Methafilcon A
Number analyzed (Participants) | 30 | 13 | 16
Number analyzed (eyes) | 60 | 26 | 32
eyes
  Grade 0 | 43 | 12 | 20
  Grade 1 | 12 | 12 | 8
  Grade 2 | 5 | 2 | 4
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

4. Primary Outcome: Bulbar Hyperemia (Redness)
Description: Subject distribution according to bulbar hyperemia scale in each eye during the 4-week Follow-up Visit. For this scale, 0 is lowest and 4 is greatest. If present in at least one eye, then it is counted.
Time Frame: 4 weeks
Population: Analysis is on those who are enrolled, randomized to a study arm, and completed the study.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Senofilcon A | Balafilcon A | Methafilcon A
Number analyzed (Participants) | 30 | 13 | 16
Number analyzed (eyes) | 60 | 26 | 32
eyes
  Grade 0 | 45 | 11 | 23
  Grade 1 | 12 | 13 | 9
  Grade 2 | 3 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

5. Primary Outcome: Corneal Staining
Description: Subject distribution according to corneal staining with fluorescein scale in each eye during the 2-week Follow-up Visit. For this scale, 0 is lowest and 4 is greatest. If present in at least one eye, then it is counted.
Time Frame: 2 weeks
Population: Analysis was on those subjects who were enrolled, randomized to a study arm, and completed the study.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Senofilcon A | Balafilcon A | Methafilcon A
Number analyzed (Participants) | 30 | 13 | 16
Number analyzed (eyes) | 60 | 26 | 32
eyes
  Grade 0 | 27 | 8 | 10
  Grade 1 | 27 | 16 | 19
  Grade 2 | 6 | 2 | 3
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

6. Primary Outcome: Corneal Staining
Description: Subject distribution according to corneal staining with fluorescein scale in each eye during the 4-week Follow-up Visit. For this scale, 0 is lowest and 4 is greatest. If present in at least one eye, then it is counted.
Time Frame: 4 weeks
Population: Analysis is on those subjects who were enrolled, randomized to a study arm, and completed the study.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Senofilcon A | Balafilcon A | Methafilcon A
Number analyzed (Participants) | 30 | 13 | 16
Number analyzed (eyes) | 60 | 26 | 32
eyes
  Grade 0 | 33 | 8 | 10
  Grade 1 | 19 | 16 | 18
  Grade 2 | 8 | 0 | 4
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Study period
Arm/Group | Senofilcon A | Lotrafilcon B | Balafilcon A | Methafilcon A | Vifilcon A
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/3 | 0/13 | 0/17 | 0/3
Other Adverse Events (participants affected / at risk) | 1/35 | 2/3 | 0/13 | 0/17 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senofilcon A (N=35) | Lotrafilcon B (N=3) | Balafilcon A (N=13) | Methafilcon A (N=17) | Vifilcon A (N=3)
Torticollis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mild Punctate Keratitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days